CLINICAL TRIAL: NCT04832464
Title: Effects of BRACE (Balance, Resistance, Aerobic and Cognitive Exercise) Protocol for Balance Training in Patients With Diabetic Peripheral Neuropathy.
Brief Title: BRACE(Balance, Resistance, Aerobic and Cognitive Exercise) Protocol for Diabetic).Peripheral Neuropathic Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00548 Azka Tariq
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: Diabetic Peripheral Neuropathy; Balance training; Strengthening; Cognitive exercises; Aerobics exercises

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training Home plan (Active Comparator): The Control group is undergoing balance training only, 3 days a week, and will be for 8 weeks. Balance training includes 10minutes of warm-up and 30 minutes of balance exercises. A force plate will be used to measure the postural sways. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
  These exercises include Static Balance exercises(1-2weeks): Romberg with eyes open & close, Tandem standing with eyes open & close with alternate feet, Single leg stance.
  Static/ Dynamic/ Anticipatory Postural Control (3-4weeks): Sit to Stand, FRT( forward reach test) that is forward, sideways, cross reach, and timed up and go test.
  Static/ Dynamic/ Anticipatory? Reactive Postural Control (5-6weeks): Perturbations:
  Controlled by the therapist in sitting & standing, Throwing a ball, kicking a ball.
  (7-8weeks): Combination of All
  Interventions: Other: RACE Protocol: Balance training along with resistance, aerobic and cognitive exercises.
- BRACE Protocol: Balance training along with resistance, aerobic and cognitive excercises (Experimental): BRACE protocol for balance training 3 days a week for 8 consecutive weeks on alternate days.
  These exercises include Static Balance exercises(1-2weeks) plus Chair rise 30 sec without using hands, 6-minute walk, count reverse from 50, push the wall, and reverse count from 20.
  Static, dynamic, anticipatory postural control (3-4weeks) plus Stair climbing without using rails, marching in space, remember 5 words, name 5 animals, repeat 5 words, spell the word like APPLE, spell backward again.
  Static, dynamic, anticipatory postural control (5-6weeks) plus Squatting, cycling, count even numbers from 1-50.
  calculation: Addition, subtraction, multiplication, division. (7-8weeks): Combination of all.
  Interventions: Other: RACE Protocol: Balance training along with resistance, aerobic and cognitive exercises.

INTERVENTIONS:
Other: RACE Protocol: Balance training along with resistance, aerobic and cognitive exercises. — therapy for the preservation, enhancement, or restoration of movement and physical function impaired or threatened by disease, injury, or disability that utilizes therapeutic exercise, physical modalities (such as massage and electrotherapy), assistive devices, and patient education and training.
  Other Names: Balance Training Home plan

SUMMARY:
The purpose of the study is to determine the effects of the BRACE( Balance, Resistance, Aerobic and Cognitive Exercise) protocol for balance training in patients with Diabetic Peripheral Neuropathy. A Randomized Control Trial is being conducted at Railways General Hospital, Rawalpindi. The sample size was calculated through the open epi tool. A total of 60 patients are divided into two groups, 30 participants in the experimental group and 30 participants in the control group. The study duration will be six months. The sampling technique applied was simple random sampling for recruitment and group randomization using the sealed envelope method. Patients with the age of 40-65 years having type II diabetes for more than 5 years are included in the study. Tools used in the study are Berg balance scale, timed up and go test, functional reach test, Montreal Cognitive Assessment scale (MOCA), and force plate. Data will be analyzed through Statistical Package for the Social Sciences (SPSS), version 21.

DETAILED DESCRIPTION:
American Diabetic Association (ADA) defined Diabetes mellitus as a group of metabolic diseases characterized by hyperglycemia resulting from defects in insulin secretion, insulin action, or both. The chronic hyperglycemia of diabetes is associated with dysfunction of various organs, especially the eyes, kidneys, nerves, heart, and blood vessels.

Most common among the neuropathies are chronic sensorimotor distal symmetric polyneuropathy (DPN) and autonomic neuropathies. According to ADA(American Diabetes Association), DPN(Diabetic Peripheral Neuropathy) is "the presence of symptoms and/or signs of peripheral nerve dysfunction in people with diabetes after exclusion of other causes. It is estimated that 60% to 70% of individuals with diabetes have mild to severe forms of nervous system damage.

DPN(Diabetic Peripheral Neuropathy) causes decreased sensation, proprioception, reflexes, and strength in the lower extremities, leading to balance dysfunction. Physical therapy interventions utilized to reduce the balance dysfunction can range from restoration of the health of the neurons to sensory integration to compensatory strategies. Various treatment protocols include improving circulation, the guided practice of integrating internal and external sensory input, education on sensation loss and fall risk, instruction on home modifications, and introduction of assistive devices to minimize balance dysfunction.

A systematic and evidence-based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines.

Search term for the initial literature review was Diabetes mellitus, the prevalence of DPN(diabetic peripheral neuropathy), causes of peripheral neuropathies and loss of balance, the pathophysiology of diabetes-related peripheral neuropathy, treatment options for balance training, strengthening lower extremities, aerobics, cognitive approach. The search was limited to papers in English preferably published since 2000 with full text available. Different studies were available regarding balance exercises and their effects but limited data was available regarding BRACE ( Balance, Resistance, Anaerobic, and Cognitive Exercise) protocol as a whole in recent years.

Balance exercises are feasible and safe and have the potential to improve balance and gait. These should be used as supportive therapy for DPN patients. Lower extremity resistance (strengthening) exercises are fairly recommended for clinical use in treating balance dysfunction in patients with DPN than monochromatic infrared energy therapy, vibrating insoles, and use of a cane.

Previously, walking and weight-bearing were considered contraindicated in DPN patients to avoid foot ulcers, deformity, or fall risk. Emerging research has revealed positive adaptations in response to overload stress in these people, including evidence for peripheral neuroplasticity in animal models and early clinical trials.

According to WHO estimation, a number of individuals approximately 47 million worldwide have cognitive impairments which will increase to 75 million by 2030. A 2 years longitudinal study in Korea showed a significant association between cognitive decline and physical activity. Pain interference may be reduced following an aerobic exercise intervention among people with painful DPN, without a change in pain intensity.

Although, multiples researches have shown the effects of particular interventions on DPN still there is a lack of multi-component interventional studies to show the effects on balance issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type-2 Diabetes
* Diabetes of more than 5 years of the duration

Exclusion Criteria:

* Patients have vertebrobasilar insufficiency (tested by VBI tests)
* Atlanto-axial instability (tested by sharp purser test)
* Osteoporosis
* Rheumatoid arthritis
* Neuropathies
* Recent surgeries

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-02-27 (Estimated); Study Completion 2022-02-27 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Up to 8 weeks
  To objectively determine a patient's ability (or inability) to safely balance during a series of pre-determined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function with a total of 56 scores. This scale is interpreted as 0-20 on the BBS represents balance impairment; 21-40 on the BBS represents acceptable balance; 41-56 on the BBS represents a good balance. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).

SECONDARY OUTCOMES:
TUG test | Up to 8 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.[1]
  It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. The scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
  Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
FRT test | Up to 8 weeks
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task. In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.
  This information is correlated with the risk of falling.
  Measurement Interpretation:
  10"/25 cm or greater Low risk of falls; 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal; 6"/15cm or less Risk of falling is 4x greater than normal; Unwilling to reach Risk of falling is 8x greater than normal. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
MoCA | Up to 8 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. In a study, people without cognitive impairment score an average of 27.4; people with mild cognitive impairment (MCI) score an average of 22.1; people with Alzheimer's disease score an average of 16.2.
  Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
Postural sway | Up to 8 weeks
  A force plate will be used to measure the postural sways. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
Gait and Posture assessment by application | Up to 8 weeks
  A mobile application (Gait and posture) will be used to measure the postural sways and balance. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).
Michigan Neuropathy Screening Instrument | Up to 8 weeks
  The Michigan Neuropathy Screening Instrument (MNSI) is designed to screen for the presence of diabetic neuropathy. The first part of the screening instrument, the history questionnaire, consists of 15 self-administered "yes or no" questions on foot sensation including pain, numbness, and temperature sensitivity. A higher score (out of a maximum of 13 points) indicates more neuropathic symptoms. The second part of the MNSI is a brief physical assessment (completed by health professionals).
  Patients screening positive on the clinical portion of the MNSI (greater than 2 points on a 10 point scale) are considered neuropathic and referred for further evaluation.
  A force plate will be used to measure the postural sways. Measurements will be taken at a base-line, after the first session, at mid-level (4th week) and at the end (8th week).

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandey S, Raj IJS. Comparison of Game Based Rehabilitation and Mixed Sport Training on Balance in Diabetic Neuropathy: Lovely Professional University; 2017
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S67-74. doi: 10.2337/dc13-S067. No abstract available. PMID 23264425
- [Background] O'Sullivan SB, Schmitz TJ, Fulk G. Physical rehabilitation: FA Davis; 2019
- [Background] Kluding PM, Bareiss SK, Hastings M, Marcus RL, Sinacore DR, Mueller MJ. Physical Training and Activity in People With Diabetic Peripheral Neuropathy: Paradigm Shift. Phys Ther. 2017 Jan 1;97(1):31-43. doi: 10.2522/ptj.20160124. PMID 27445060
- [Background] Ahmad I, Hussain E, Singla D, Verma S, Ali K. Balance Training in Diabetic Peripheral Neuropathy: A Narrative Review. JSM Diabetol Manag. 2017;2(1):1-9
- [Background] Wallin A, Kettunen P, Johansson PM, Jonsdottir IH, Nilsson C, Nilsson M, Eckerstrom M, Nordlund A, Nyberg L, Sunnerhagen KS, Svensson J, Terzis B, Wahlund LO, Georg Kuhn H. Cognitive medicine - a new approach in health care science. BMC Psychiatry. 2018 Feb 8;18(1):42. doi: 10.1186/s12888-018-1615-0. PMID 29422020
- [Background] Kiani N, Marryam M, Malik AN, Amjad I. The effect of aerobic exercises on balance in diabetic neuropathy patients. Journal Of Medical Sciences. 2018;26(2):141-5